CLINICAL TRIAL: NCT06452277
Title: A Phase 3 Open-label, Randomized, Active-controlled, Multicenter Trial to Evaluate the Efficacy and Safety of Orally Administered BAY 2927088 Compared With Standard of Care as a First-line Therapy in Patients With Locally Advanced or Metastatic Non-small Cell Lung Cancer (NSCLC) With HER2-activating Mutations
Brief Title: A Study to Learn More About How Well Sevabertinib (BAY 2927088) Works and How Safe it is Compared With Standard Treatment, in Participants Who Have Advanced Non-small Cell Lung Cancer (NSCLC) With Mutations of the Human Epidermal Growth Factor Receptor 2 (HER2)
Acronym: SOHO-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22615; 2024-511319-91-00 (Other: CTIS (EU))
Expanded Access: NCT06761976 (Available)
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Advanced Non-small Cell Lung Cancer; HER2 Mutation
Keywords: NSCLC; ERBB2 mutation
MeSH Terms: interventions — pembrolizumab; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BAY2927088 (Experimental): Participants will receive BAY2927088 20 mg BID until disease progression per RECIST v1.1, unacceptable toxicity, or until any other withdrawal criteria.
  Interventions: Drug: BAY2927088
- Standard of care (SoC) (Active Comparator): Participants will receive SoC (pembrolizumab in combination with platinum-based chemotherapy, in 21-day cycles per the approved labels) until disease progression per RECIST v1.1, unacceptable toxicity, or until any other withdrawal criteria.
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: BAY2927088 — Tablet, oral
  Arms: BAY2927088
Drug: Pembrolizumab — Intravenous (IV) infusion
  Arms: Standard of care (SoC)
Drug: Cisplatin — IV infusion
  Arms: Standard of care (SoC)
Drug: Carboplatin — IV infusion
  Arms: Standard of care (SoC)
Drug: Pemetrexed — IV infusion
  Arms: Standard of care (SoC)

SUMMARY:
Researchers are looking for a better way to treat people who have advanced non-small cell lung cancer (NSCLC) with specific genetic changes called human epidermal growth factor receptor 2 (HER2) mutations.

Advanced NSCLC is a group of lung cancers that have spread to nearby tissues or to other parts of the body or that are unlikely to be cured or controlled with currently available treatments. HER2 is a protein that helps cells to grow and divide. A damage (also called mutation) to the building plans (genes) for this protein in cancer cells leads to a production of abnormal HER2 and therefore abnormal cell growth and division.

The study treatment, BAY 2927088, is expected to block the mutated HER2 protein which may stop the spread of NSCLC.

The main purpose of this study is to learn how well BAY 2927088 works and how safe it is compared with standard treatment, in participants who have advanced NSCLC with specific genetic changes called HER2 mutations.

The study participants will receive one of the study treatments:

* BAY 2927088 twice every day as a tablet by mouth, or
* Standard treatment in cycles of 21 days via infusion ("drip") into the vein. The treatment will continue for as long as participants benefit from it without any severe side effects or until they or their doctor decide to stop the treatment.

During the study, the doctors and their study team will:

* take imaging scans, including CT, PET, MRI, and X-rays, of different parts of the body to study the spread of cancer
* check the overall health of the participants by performing tests such as blood and urine tests, and checking
* heart health using an electrocardiogram (ECG)
* perform pregnancy tests for women
* ask the participants questions about how they are feeling and what adverse events they are having.

An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events, irrespective if they think it is related or not to the study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age or over the legal age of consent in countries where that is greater than 18 years at the time of signing the informed consent.
* Documented histologically or cytologically confirmed locally advanced non-squamous NSCLC, not suitable for definitive therapy or metastatic non-squamous NSCLC at screening (small cell or mixed histologies are excluded) (Stage III-IV NSCLC).
* Documented activating HER2 mutation in the tyrosine kinase domain (TKD) assessed by tissue molecular test in a CLIA-certified (US sites) or an equally accredited (outside of the US) local laboratory. However, participants may be included at the discretion of the investigator if the laboratory performing the assay is not CLIA or similar certified but the laboratory is locally accredited.
* No prior systemic therapy for locally advanced or metastatic disease. No prior treatment with a HER2 ex20ins-targeted therapy (e.g. poziotinib, trastuzumab deruxtecan). Participants who received adjuvant or neoadjuvant therapy are eligible if the adjuvant/neoadjuvant therapy was completed at least 12 months prior to the start of screening.
* Eligible to receive treatment with the selected platinum-based doublet-chemotherapy (i.e. cisplatin/pemetrexed or carboplatin/pemetrexed) and pembrolizumab in accordance with the SmPC/Product Information.

Exclusion Criteria:

* Known history of prior malignancy except if the participant has undergone potentially curative therapy with no evidence of that disease recurrence for five years since initiation of that therapy. Exception: the following cancer types are acceptable within five years if curatively treated or under surveillance:

  * a. in situ cancers of cervix, breast, or skin,
  * b. superficial bladder cancer (Ta, Tis and T1),
  * c. limited-stage prostate cancer,
  * d. basal or squamous cancers of the skin.
* Tumors with targetable alterations with approved available therapy, with the exception of HER2 mutation in the TKD.
* Inability to discontinue treatment with chronic systemic corticosteroids. Participants who require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study. Replacement therapy (e.g., physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is acceptable, provided that the dose is stable for >4 weeks prior to planned start of study intervention.
* Pre-existing peripheral neuropathy that is Grade ≥2 by CTCAE (v5.0).
* History of severe hypersensitivity reaction to treatment with a monoclonal antibody.
* Prior radiotherapy outside of the brain within 21 days before of planned start of study intervention. Participants must have recovered from all radiation-related toxicities and not require corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-10-28 (Estimated); Study Completion 2029-06-27 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) per RECIST 1.1 as assessed by BICR | Up to approximately 2 years
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; BICR = blinded independent central review (BICR)

SECONDARY OUTCOMES:
Overall survival (OS) | Up to approximately 4 years.
Objective response rate (ORR) per RECIST 1.1 as assessed by BICR | Up to approximately 4 years
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; BICR = blinded independent central review (BICR)
Progression free survival (PFS) per RECIST 1.1 as assessed by the investigator | Up to approximately 4 years
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1
Objective Response Rate (ORR) per RECIST 1.1 as assessed by the investigator | Up to approximately 4 years
Disease control rate (DCR) per RECIST 1.1 as assessed by BICR | Up to approximately 4 years
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1; BICR = blinded independent central review (BICR)
Disease control rate (DCR) per RECIST 1.1 as assessed by the investigator | Up to approximately 4 years
  RECIST 1.1 = Response Evaluation Criteria in Solid Tumors, version 1.1
Duration of response (DOR) as assessed by BICR | Up to approximately 4 years
  BICR = blinded independent central review (BICR)
Duration of response (DOR) as assessed by the investigator | Up to approximately 4 years
Adverse events per CTCAE v 5.0 (eg. TEAEs, TESAEs) categorized by severity | Up to approximately 4 years
  CTCAE = common terminology criteria for adverse events; TEAE = treatment-emergent adverse event; TESAE = treatment-emergent serious adverse event
Change from baseline in NSCLC-SAQ total score | Up to approximately 4 years
  NSCLC-SAQ = Non-small cell lung cancer Symptom Assessment Questionnaire
Change from baseline in NSCLC-SAQ individual domain scores | Up to approximately 4 years
  NSCLC-SAQ = Non-small cell lung cancer Symptom Assessment Questionnaire; Domains: cough, pain, dyspnea, fatigue, appetite
Time to deterioration in NSCLC-SAQ total score | Up to approximately 4 years
  NSCLC-SAQ = Non-small cell lung cancer Symptom Assessment Questionnaire
Time to deterioration in NSCLC-SAQ individual domain scores | Up to approximately 4 years
  NSCLC-SAQ = Non-small cell lung cancer Symptom Assessment Questionnaire; Domains: cough, pain, dyspnea, fatigue, appetite
Time to deterioration in EORTC QLQ-C30 physical functioning domain score | Up to approximately 4 years
  EORTC QLQ-C30: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30
Change from baseline in EORTC QLQ-C30 physical functioning domain score | Up to approximately 4 years
  EORTC QLQ-C30: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30; QoL: quality of life
Change from baseline in EORTC QLQ-C30 global health status/QoL | Up to approximately 4 years
  EORTC QLQ-C30: European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30; QoL: quality of life

CONTACTS AND LOCATIONS:
Locations (278):
- United States (26):
  - Patty & George Hoag Cancer Center, Newport Beach, California
  - UC San Diego Health - Moores Cancer Center, San Diego, California
  - UCSF Bakar Precision Cancer Medicine Building - Thoracic Surgery and Oncology, San Francisco, California
  - UCLA Health Santa Monica Cancer Care, Santa Monica, California
  - The Oncology Institute of Hope and Innovation - Fort Lauderdale 17th Street, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Miramar, Miramar, Florida
  - AdventHealth Cancer Institute Orlando, Orlando, Florida
  - Moffitt Cancer Center - Magnolia Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Piedmont Cancer Institute - Atlanta, Atlanta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - University of Illinois Hospital - Outpatient Cancer Care Center, Chicago, Illinois
  - The University of Chicago Medical Center - Hyde Park - Hematology & Oncology, Chicago, Illinois
  - UM Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - UMass Memorial Medical Center - University Campus - Hematology/Oncology, Worcester, Massachusetts
  - Profound Research -OMG - TriAtria Cancer Center, Farmington Hills, Michigan
  - Profound Research - OMG - Royal Oak Cancer Center, Royal Oak, Michigan
  - M Health Fairview Masonic Cancer Clinic - Clinics and Surgery Center, Minneapolis, Minnesota
  - R.J. Zuckerberg Cancer Center, New Hyde Park, New York
  - UC Medical Center - Oncology, Cincinnati, Ohio
  - Providence Cancer Institute - Franz Clinic, Portland, Oregon
  - Providence Oncology and Hematology Care Clinic Westside, Portland, Oregon
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University Hospital Simmons Cancer Center Lung/Head Neck Clinic, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center - Texas Medical Center, Houston, Texas
  - VCU Health Ambulatory Care Center - Cardiology, Richmond, Virginia
- Argentina (6):
  - Fundación Cenit para la Investigación en Neurociencias, CABA, Ciudad Auton. de Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Centro de Educacion Medica e Investigaciones Clinicas "Norberto Quirno" (CEMIC), Buenos Aires
  - Centro Médico Privado CEMAIC, Córdoba
  - Instituto Argentino de Diagnostico y Tratamiento (IADT), TBC
  - Centro de Investigaciones Clínicas, Clínica Viedma, Viedma
- Australia (6):
  - NSW Health - Blacktown Hospital, Blacktown, New South Wales
  - Concord Repatriation General Hospital - Medical Oncology Clinical Trials Unit, Concord, New South Wales
  - Calvary Mater Hospital Newcastle - Oncology, Waratah, New South Wales
  - University of the Sunshine Coast, Buderim, Queensland
  - Austin Hospital - Olivia Newton John Cancer Research Institute, Heidelberg, Victoria
  - The Canberra Hospital (TCH) - Canberra Region Cancer Centre (CRCC), Garran
- Austria (4):
  - Uniklinikum Salzburg, Universitätsklinik für Innere Medizin III, Vienna, Salzburg
  - Uniklinikum Salzburg, Universitätsklinik für Pneumologie/ Lungenheilkunde, Vienna, Salzburg
  - Medizinische Universität Wien Universitätsklinik f. Innere Medizin I Klinische Abteilung für Onkologie, Vienna, Vienna
  - Klinik Floridsdorf, Pneumo-onkologische Ambulanz und Tagesklinik, Vienna
- Belgium (3):
  - UZ Leuven Gasthuisberg - Pneumology Department, Leuven, Vlaams-Brabant
  - AZ Delta | Clinical Trial Center - Pneumology, Roeselare, West-Flanders
  - Antwerp University Hospital | Oncology Department, Antwerp
- Brazil (12):
  - Rede DoR Recife - PE, Recife, Pernambuco
  - Liga Norte Riograndense Contra o Cancer | Centro de Pesquisa Clínica, Natal, Rio Grande do Norte
  - Irmandade Santa Casa de Misericordia de Porto Alegre | Oncology, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa da Clínica de Oncologia Reichow, Blumenau, Santa Catarina
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital de Base | Funfarme - Centro Integrado de Pesquisa - Cardiologia, São José do Rio Preto, São Paulo
  - NAIC - Instituto do Cancer, Bauru
  - Hospital Sirio-Libanes (HSL) - Centro de Oncologia - Brasilia, Brasília
  - Pronutrir Fortaleza - CE, Fortaleza
  - Hospital Sirio Libanes, São Paulo
  - A Beneficencia Portuguesa de Sao Paulo - Hospital BP Mirante, São Paulo
  - Centro Paulista de Oncologia (CPO) - Sao Paulo - Faria Lima, São Paulo
- Bulgaria (9):
  - MHAT Uni Hospital, Panagyurishte, Pazardzhik
  - MHAT "Heart and brain" Pleven, Pleven
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - MHAT Park Hospital EOOD, Plovdiv
  - Multiprofile Hospital for Active Treatment "Sveta Sofia", Sofia
  - MHAT Serdika, Sofia
  - Specialized Hospital for Active Treatment of Oncology, Sofia
  - University Multiprofile Hospital For Active Treatment Sofiamed OOD, Sofia, Sofia
  - MHAT Sveta Marina EAD, Varna
- Canada (4):
  - BC Cancer - Vancouver Site, Vancouver, British Columbia
  - Brampton Civic Hospital - Oncology, Brampton, Ontario
  - Princess Margaret Cancer Centre - University Health Network - Department of Medical Oncology and Hematology, Toronto, Ontario
  - Jewish General Hospital - Department of Pulmonary Oncology, Montreal, Quebec
- China (25):
  - Beijing Cancer Hospital - Oncology Department, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Union Hospi, Tongji Med College, Huazhong Univ. Scien&Tech, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital - Oncology Department, Changsha, Hunan
  - NJ Drum Tower Hospital, the Affil Hos of NJ Univ Med School, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Shanghai Chest Hospital, Shanghai Jiaotong University, Shanghai, Shanghai Municipality
  - West China Hospital Sichuan University, Chengdu, Sichuan
  - Sir Run Run Shaw Hospital, Zhejiang Univ. School of Medicine - Oncology Department, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Zhejiang University School of Medicine - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - The People's Liberation Army General Hospital (Beijing 301 Hospital), Beijing
  - Beijing chest hospital, Capital Medical University, Beijing
  - University of Electronic Science & Technology of China - Sichuan Cancer Hospital & Institute (Sichuan Provincial Tumor Hospital), Chengdu
  - Guangzhou Medical University - The First Affiliated Hospital, Guangzhou
  - Shandong University - Shandong Cancer Hospital, Jinan
  - LinYi Cancer Hospital (Linyi Tumor Hospital), Linyi
  - Jiangsu Provincial People's Hospital - The First Affiliated Hospital of Nanjing Medical University, Nanjing
  - Guangxi Medical University (GXMU) - Affiliated Tumor Hospital, Nanning
  - Zhongshan Hospital, Fudan University - Oncology Department, Shanghai
  - Xiamen University - The First Affiliated Hospital, Xiamen
- Czechia (5):
  - Krajská nemocnice T. Bati - Pneumoonkologická a klinická onkologie, Zlín, Zlín
  - Masarykova Univerzita - Masarykuv Onkologicky Ustav (MOU) - Klinika Komplexni Onkologicke Pece (KKOP), Brno
  - Nemocnice AGEL Nový Jicín a.s. - Oddelení radioterapie a onkologie, Nový Jicín
  - Fakultní Nemocnice Olomouc - Klinika plicních nemocí a tuberkulózy, Olomouc
  - Nemocnice AGEL Ostrava-Vítkovice a. s. - Plicní oddelení, Ostrava - Vítkovice
- Denmark (5):
  - Aalborg University hospital - oncology department, Aalborg
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet - Kræftbehandling, Copenhagen OE
  - Regionshospitalet Gødstrup - Medicinsk afdeling, Herning
  - Odense University Hospital - Oncology Department, Odense C
- Finland (2):
  - Docrates Mehiläinen Syöpäsairaala, Helsinki, Uusimaa
  - Turku University Hospital, Turun yliopistollinen sairaala (TYKS) - Keuhkosairauksien poliklinikka, Turku
- France (17):
  - Institut Bergonie - Unicancer Nouvelle Aquitaine, Bordeaux
  - Hopital La Cavale Blanche - CHU de Brest - institut de cancerologie et d'imagerie, Brest
  - Centre Hospitalier Intercommunal Creteil - Service de pneumologie, Créteil
  - Centre Hospitalier Michallon Grenoble - Service pneumologie, La Tronche
  - Institut Coeur Poumon CHRU Lille - Pole Cardio-vasculaire et pulmonaire, Lille
  - Centre Hospitalier Universitaire de Limoges - unite oncologie thoracique, Limoges
  - CHU Montpellier - Hopital Arnaud de Villeneuve - Service oncologie thoracique, Montpellier
  - hopital Emile Muller - Service Pneumologie, Mulhouse
  - Hopital Nord Laennec - Oncologie medicale thoracique et digestive, Nantes
  - Centre Antoine Lacassagne - Departement Oncologie, Nice
  - hopital cochin APHP - service de pneumologie, Paris
  - Institut Curie - Paris - Oncologie medicale, Paris
  - hopital Lyon sud HCL - Pneumologie aigue specialisee et cancerologie thoracique, Pierre-Bénite
  - CHU de Rouen - Hopital Charles Nicolle - Service de Pneumologie, Rouen
  - Institut de Cancerologie Ouest - Saint-Herblain, Saint-Herblain
  - Hopital Foch - Oncologie digestive et thoracique, Suresnes
  - Gustave Roussy - Departement Oncologie-Radiotherapie, Villejuif
- Germany (8):
  - Universitaetsklinikum Giessen und Marburg - Medizinische Klinik IV Organonkologie, Giessen, Hesse
  - Kliniken der Stadt Köln gGmbH - Krankenhaus Merheim - Lungenklinik, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Essen - Innere Klinik (Tumorforschung), Essen, North Rhine-Westphalia
  - Charité Universitätsmedizin Berlin CBF - Med. Klinik mit Schwerpunkt Hämatologie, Onkologie und Tumorimmunologie, Berlin
  - Universitätsklinikum Frankfurt - Medizinische Klinik II, Hämatologie und Onkologie, Frankfurt
  - Lungenklinik Hemer, Thorakale Onkologie und onkologische Palliativmedizin, Hemer
  - Klinikum Nürnberg - Klinik für Innere Medizin 3, Schwerpunkt Pneumologie (Lungenheilkunde), Nuremberg
  - Robert Bosch Krankenhaus - Haematologie, Onkologie und Palliativmedizin, Stuttgart
- Greece (9):
  - General University Hospital Of Larissa-Department of Medical Oncology, Mezourlo, Larisa
  - Henry Durant Hospital Center-4th Oncology Department and Clinical Trials Unit, Athens
  - Thoracic General Hospital Of Athens I Sotiria-3rd University Department of Internal Medicine, Athens
  - General Hospital of Athens "Alexandra''-Plasma Cell Dyscrasias,Department of Clinical Therapeutics,School of Medicine,NKUA, Athens
  - University General Hospital Attikon, 2nd Department of Propaedeutic and Internal Medicine, Athens
  - University General Hospital Attikon-4th Department of Internal Medicine, Chaïdári
  - Metropolitan Hospital- 4th Oncology Clinic, Piraeus
  - Bioclinic Thessaloniki, Thessaloniki
  - Geniko Nosokomeio Thessalonikis George Papanikolaou-Pulmonary Department, Thessaloniki
- Hong Kong (4):
  - Prince of Wales Hospital, Hong Kong, Hong Kong SAR
  - Queen Elizabeth Hospital Hong Kong, Hong Kong, Hong Kong SAR
  - Queen Mary Hospital, Hong Kong, Hong Kong SAR
  - Hong Kong United Oncology Centre, Kowloon
- Hungary (2):
  - Budapesti Uzsoki Utcai Korhaz - Tüdogyógyászati Osztály, Budapest
  - Komarom-Esztergom Varmegyei Szent Borbala Korhaz, Tatabánya
- Israel (4):
  - Assuta Ashdod Public Hospital (R.A), Ashdod
  - Soroka Medical Center- Legacy Heritage Cancer Center, Beersheba
  - Shaare Zedek Medical Center (SZMC), Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (17):
  - AORN San Giuseppe Moscati Avellino - U.O.C. Oncologia Medica, Avellino, Campania
  - Azienda Ospedaliero-Universitaria Di Bologna IRCCS_Policlinico Sant'Orsola - UOC Oncologia Medica, Bologna, Emilia-Romagna
  - Istituto Romagnolo Per Lo Studio Dei Tumori Dino Amadori IRST S.r.l. - GDP Toracica, Meldola, Emilia-Romagna
  - Centro di Riferimento Oncologico di Aviano - Oncologia Medica e dei Tumori Immuno-Correlati, Aviano, Friuli Venezia Giulia
  - I.F.O. Istituti Fisioterapici Ospitalieri_Ospedale Regina Elena -- Oncologia Medica 2, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOSD Oncologia Toraco-Polmonare, Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori - S. C. Oncologia Medica 1, Milan, Lombardy
  - Istituto Europeo di Oncologia s.r.l - Oncologia Toracica, Milan, Lombardy
  - Humanitas Mirasole S.p.A. - Oncologia Medica ed Ematologia, Rozzano, Lombardy
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga - Oncologia Medica, Orbassano, Piedmont
  - Istituto Oncologico Veneto_Padova - UOC Oncologia 2, Padua, Veneto
  - Careggi University Hospital - Oncologia Clinica, Florence
  - Ospedale Vito Fazzi Lecce - Oncologia, Lecce
  - Ospedale San Raffaele s.r.l. - Oncologia Medica, Milan
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello - Oncologia Medica, Palermo
  - ASST Sette Laghi_Ospedale Macchi - Oncologia, Varese
  - Centro Ricerche Cliniche Di Verona S.r.l. - Oncologia, Verona
- Japan (16):
  - National Hospital Organization Nagoya Medical Center, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - National Hospital Organization Himeji Medical Center, Himeji, Hyōgo
  - Kobe University Hospital, Kobe, Hyōgo
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital, Sakai, Osaka
  - Saitama Cancer Center, Kitaadachi-gun, Saitama
  - Nippon Medical School - Nippon Medical School Hospital - Cancer Center, Bunkyo-ku, Tokyo
  - Tottori University Hospital, Yonago, Tottori
  - National Hospital Organization-Yamaguchi-Ube Medical Center (Sanyo Hospital), Ube, Yamaguchi
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Niigata Cancer Center Hospital, Niigata
  - Osaka International Cancer Institute, Osaka
- Malaysia (7):
  - Beacon Hospital, Petaling Jaya, Selangor
  - Columbia Asia Hospital Bukit Rimau, Shah Alam, Selangor
  - Sunway Medical Centre, Subang Jaya, Selangor
  - University Hospital Kebangsaan Malaysia, Cheras
  - Gleneagles Penang Medical Center, George Town
  - Universiti Malaya Medical Centre, Kuala Lumpur
  - Sunway Medical Centre Penang, Perai
- Mexico (6):
  - Instituto Nacional de Cancerología, Mexico City, Mexico City
  - Oncare Viaducto Nápoles, Mexico City
  - Oncología Integral Satélite, Naucalpan
  - Hospital Universitrio Dr. José Eleuterio González. Servicio de Oncologia, Nuevo León
  - Clinica Integral Internacional de Oncologia S. de R.L. de C.V., Puebla City
  - ONCARE Treatment Center, San Pedro Garza García
- Netherlands (2):
  - Nederlands Kanker Instituut, Amsterdam
  - Radboud University Medical Center | Afdeling Interne Geneeskunde, Nijmegen
- Poland (8):
  - Narodowy Instytut Onkologii-im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy - Nowotworow Pluca i Klatki Piersiowej, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Swietokrzyskie Centrum Onkologii, Kielce
  - Uniwersytecki Szpital Kliniczny Nr 2 Uniwersytetu Medycznego w Lodzi, Lodz
  - Mazowieckie Centrum Leczenia Chorob Pluc i Gruzlicy w Otwocku, Otwock
  - Wielkopolskie Centrum Pulmonologii i Torakochirurgii, Poznan
  - Instytut Gruzlicy i Chorob Pluc, Warsaw
  - Dolnoslaskie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw
- Portugal (5):
  - Hospital Pedro Hispano | Clinical Research Center, Matosinhos Municipality, Porto District
  - Unidade Local Saúde Coimbra, E.P.E, Coimbra
  - Fundacao Champalimaud | Centro Clinico Champalimaud - Unidade Investigacao Clinica, Lisbon
  - CHULN - Hospital Pulido Valente, Lisbon
  - IPO Porto, Porto
- Romania (9):
  - Radiotherapy Center Cluj SRL, Flore?ti, Comuna Floresti
  - Institutul Oncologic Prof. Dr. Alexandru Trestioreanu (IOB); Oncologie Medicala II, Bucharest
  - Spitalul Clinic Coltea, Bucharest
  - CardioMed S.R.L., Cluj-Napoca
  - Institutul Oncologic Prof. Dr. Ion Chiricuta, Cluj-Napoca
  - Sc Oncolab Srl, Craiova
  - Centrul de Oncologie Sfantul Nectarie, Craiova
  - S.C Ovidius Clinical Hospital SRL - Oncology Department, Ovidiu
  - Oncocenter, Timișoara
- Singapore (4):
  - Raffles Cancer Centre, Singapore
  - OncoCare Cancer Centre | Gleneagles Medical Centre, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Curie Oncology | Farrer, Singapore
- Slovakia (2):
  - POKO Poprad s.r.o., Poprad
  - Fakultna nemocnica Trnava, Trnava
- South Korea (7):
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Severance Hospital, Yonsei University Health System - Oncology Department, Seoul, Seoul Teugbyeolsi
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi
  - Chonnam National University Hwasun Hospital | Pulmonology and Critical Care Medicine, Hwasun Gun
  - Samsung Medical Center - Oncology Department, Seoul
- Spain (12):
  - Hospital Germans Trias I Pujol | Oncologia, Badalona, Barcelona
  - Hospital Universitario Puerta De Hierro De Majadahonda | Oncologia, Majadahonda, Madrid
  - Hospital Universitario De Navarra | Oncologia, Pamplona, Navarre
  - Complexo Hospitalario Universitario A Coruna | Oncologia, A Coruña
  - Hospital Universitari Dexeus Grupo Quironsalud | Oncologia, Barcelona
  - Hospital Universitari Vall D Hebron | Oncologia, Barcelona
  - Hospital Clinic De Barcelona | Oncologia, Barcelona
  - Hospital General Universitario Gregorio Maranon | Oncologia, Madrid
  - Hospital Universitario Ramon Y Cajal | Oncologia, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz | Oncologia, Madrid
  - Fundacion Instituto Valenciano De Oncologia | Oncologia, Valencia
  - Hospital Universitario Y Politecnico La Fe | Oncologia, Valencia
- Sweden (2):
  - Skåne University Hospital, Lund
  - Norrland University Hospital - Cancercentrum, Umeå
- Switzerland (2):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - HFR Freiburg - Kantonsspital, Fribourg
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Kaohsiung
  - National Cheng Kung University Hospital, Tainan, TNN
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi-Mei Medical Center, Liouyine, Tainan
  - National Taiwan University Hospital (NTUH) - Cancer Research Center, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Turkey (Türkiye) (8):
  - Adana Sehir Egitim ve Arastirma Hastanesi, Yüreğir, Adana
  - Ankara Bilkent Sehir Hastanesi, Bilkent Ankara, Ankara
  - Ankara Etlik Sehir Hastanesi, Yenimahalle, Ankara
  - Istanbul Medeniyet Üniversitesi Göztepe Süleyman Yalçin Sehir Hastanesi, Kadıköy, Istanbul
  - I.A.Ü. VM Medical Park Florya Hastanesi, Küçükçekmece, Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi, Istanbul
  - Ege Universitesi Tip Fakultesi Hastanesi, Izmir
  - Sakarya Universitesi Egitim ve Arastirma Hastanesi, Sakarya
- Ukraine (8):
  - LLC "RDP Ukraine" - Medical Department, Dnipro
  - Private Enterprise Private Production Company "Acinus", Treatment and Diagnostic Center, Kropyvnytskyi
  - Kyiv City Clinical Oncology Center - Department of Chemotherapy #1, Kyiv
  - Limited Liability Company "MedOffice Group Medical Center", Kyiv
  - Medical Center LLC "Verum Expert Clinic", Kyiv
  - Volyn Regional Oncology Center, Lutsk
  - Municipal Enterprise Rivne Regional Antitumor Center of the Rivne Regional Council, Abdominal department, Rivne
  - MNCE "Uzhhorod City Multidisciplinary Clinical Hospital" -Oncology Department, Uzhhorod
- United Kingdom (4):
  - Torbay Hospital, Torquay, Devon
  - Belfast City Hospital, Belfast, Northern Ireland
  - Royal Surrey County Hospital, Guildford, Surrey
  - Velindre University NHS Trust | Velindre Cancer Centre - Clinical Trials Unit, Cardiff, Wales

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22615